CLINICAL TRIAL: NCT01602484
Title: Application Time of Plaster-of-Paris Splint Packs Compared to Bulk Supplies Following Standard Orthopaedic Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Eric Bluman, Research Director, Brigham Foot and Ankle Clinic, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2011P002091
Record Dates: First submitted 2012-05-16; First posted 2012-05-21 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Post-operative Time Saving Techniques

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Splint Pack (Experimental): Group of post-op patients who have splint applied from prepared Plaster-of-Paris splint pack
  Interventions: Device: Pre-prepared Splint Pack composed by Medline
- Bulk Supplies (Active Comparator): Group of post-op patients who have splint applied from bulk supplies
  Interventions: Device: Bulk splint supplies

INTERVENTIONS:
Device: Pre-prepared Splint Pack composed by Medline — Applying splint by using pre-prepared splint pack
  Arms: Splint Pack
Device: Bulk splint supplies — Applying splint by using the bulk splint supplies
  Other Names: Standard supplies used to create post-op splint
  Arms: Bulk Supplies

SUMMARY:
The investigators wish to perform a randomized controlled study to determine how much time and money is saved by orthopedic foot and ankle surgeons through the use of prepared splint packs compared to bulk supplies.

DETAILED DESCRIPTION:
The most expensive variable in the operating room (OR) is time. At the Faulkner hospital one hour of OR time costs approximately $500, exclusive of supply and personnel costs. Many things contribute to the amount of time a surgical procedure takes. One of these is application of the post surgical immobilization required of almost all orthopedic surgery cases. Custom molded Plaster-of-Paris splints are used for immobilization after the vast majority of orthopedic foot and ankle procedures. They have many advantages including exact fit for each patient, low cost and excellent safety profile. Traditionally these splints are constructed from bulk supplies at the end of surgical cases. The collection, measurement and organization of the component materials require the circulating nurse or surgeon to devote time to these tasks. This necessarily precludes OR staff from performing other tasks in the OR and lengthens the overall case duration. By lengthening the duration of the case more cost is incurred. The total number of cases able to be completed in a single operative day may also be diminished by the aggregate increased case time. Recently, the investigators have started utilizing prepared splint packs containing all components necessary for single plaster-of-Paris splint applications. This alternative to the traditional method of splint application has minimal expense over that incurred with traditional methods. Pilot studies have shown that the use of these splint packs diminish the time of application by 50 percent.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing post-operative standard Plaster-of-Paris splint application

Exclusion Criteria:

* amputation of foot or lower limb,
* procedure limited to skin or removal of superficial hardware,
* BMI ≥ 40,
* a medical condition that is contraindication for splint application, or
* an allergy to Plaster-of-Paris

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Bluman, M.D., Ph.D., Principal Investigator — Brigham Foot and Ankle Clinic
Locations (1):
- Faulkner Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During a six-month period from November 2011 to May 2012, fifty patients met inclusion criteria, 29 females and 21 males. Twenty-five patients were randomized to each group. The subjects were patients of the Brigham Foot and Ankle Clinic and had surgery performed at Faulkner Hospital in Boston, MA.
Pre-assignment Details: No enrolled patients were excluded from study or excluded from assignment to groups.
Period: Overall Study
Arm/Group | Splint Pack | Bulk Supplies
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Not completed — Airway issues unrelated to study | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Splint Pack | Bulk Supplies | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 16 | 19 | 35
  >=65 years | 8 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.45 (18.41) | 56.30 (16.81) | 56.37 (17.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Total Splint Application Time
Description: Time it takes to apply post-op splint
Time Frame: Immediately following the operation, beginning at the start of gathering splint supplies and ending when splint application is completed (approximately five total minutes)
Population: One patient from the bulk supply group because the subject's splinting was interrupted secondary to airway issues not related to the study.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Splint Pack | Bulk Supplies
Number analyzed (Participants) | 25 | 24
seconds | 354 [341 to 368] | 526 [512 to 541]

2. Secondary Outcome: Time to Gather Supplies
Description: Time it takes to gather supplies prior to splint application
Time Frame: Immediately following the operation, beginning with when medical personnel start to gather supplies and ending when they finish gathering supplies (approximately 1 minute)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Splint Pack | Bulk Supplies
Number analyzed (Participants) | 25 | 24
seconds | 33 [29 to 37] | 68 [61 to 76]

3. Secondary Outcome: Time to Prepare Splint
Description: Time it takes to prepare splint supplies prior to splint application
Time Frame: Immediately following the operation, beginning with when medical personnel finish gathering supplies and ending when the materials are prepared to apply splint (approximately 2 minutes)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Splint Pack | Bulk Supplies
Number analyzed (Participants) | 25 | 24
seconds | 86 [80 to 92] | 209 [198 to 220]

4. Secondary Outcome: Time to Apply Splint
Description: Time it takes to apply splint
Time Frame: Immediately following the operation, beginning with when medical personnel finish preparing supplies and ending when the splint is applied (approximately 3 minutes)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Splint Pack | Bulk Supplies
Number analyzed (Participants) | 25 | 24
seconds | 235 [227 to 244] | 249 [238 to 261]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Splint Pack | Bulk Supplies
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Splinting for one patient was interrupted secondary to airway issues unrelated to the study, so this subject was excluded from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No